CLINICAL TRIAL: NCT01799330
Title: Rehabilitation of Patients With COPD Using Electrical Muscle Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0809004250
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: COPD
Keywords: COPD; Rehabilitation; Exercise; TCEMS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1:Active TCEMS (Experimental): Transcutaneous Electrical Muscle Stimulation (TCEMS): Group 1 will undergo TCEMS using an Omnistim FX-2 with two surface patch electrodes (8 x 6 cm) applied to each quadriceps, hamstring and calf muscles. The knee angle will remain at 90 degrees during simultaneous muscle stimulation to prevent joint movement. Electrical stimulation will be performed for 20 minutes on each limb, 3 days/week for 8 continuous weeks on an outpatient basis. The stimulator will be set to generate brief bursts of electrical impulses at 50Hz lasting 200 ms every 1500 ms. Muscles will be stimulated with an asymmetrical square wave pulse with an initial intensity set to create a visible contraction ranging from 55 mA to 120 mA.
  Interventions: Procedure: Transcutaneous Electrical Muscle Stimulation (TCEMS)
- Group 2: Sham TCEMS (Placebo Comparator): Patients randomized to Group 2 (Sham TCEMS) will receive the identical set-up for active TCEMS except they will receive a minimal electrical stimulus that does not produce a motor response.
  Interventions: Other: Sham TCEMS

INTERVENTIONS:
Procedure: Transcutaneous Electrical Muscle Stimulation (TCEMS)
  Arms: Group 1:Active TCEMS
Other: Sham TCEMS — Patients randomized to Group 2 (Sham TCEMS) will receive the identical set-up for active TCEMS except they will receive a minimal electrical stimulus that does not produce a motor response
  Arms: Group 2: Sham TCEMS

SUMMARY:
The two hypotheses to be tested in this study are that:

1. The administration of transcutaneous electrical muscle stimulation (TCEMS) after completion of conventional exercise training in pulmonary rehabilitation (PR) will result in further improvements in exercise tolerance, functional status and symptoms of patients with stable chronic obstructive pulmonary disease (COPD) above those achieved in PR alone.
2. TCEMS can improve exercise tolerance, functional status and symptoms even among COPD patients who fail to make gains in exercise tolerance by participating in conventional PR due to their debilitation and/or marked cardio-respiratory impairment.

DETAILED DESCRIPTION:
Although a substantial body of evidence supports the existence of skeletal muscle dysfunction in COPD and the benefits of PR for these patients, the role of TCEMS as a routine rehabilitative strategy for patients with COPD has yet to be established. The studies proposed in this research will build on the knowledge gained in our previous study of TCEMS by investigating whether and how TCEMS adds to the beneficial effects of PR on exercise capacity and muscle function among outpatients with stable COPD, and by assessing for the first time whether TCEMS improves exercise tolerance and functional status among COPD patients unable to make gains following conventional outpatient PR. Thus, this proposed study may provide a novel strategy in the rehabilitation of patients with chronic lung disease.

The two specific aims of the proposed study are:

1. Determine whether administration of TCEMS after conventional exercise training in PR leads to added gains in muscle strength, exercise capacity, dyspnea and health status, to determine if TCEMS should be considered as an additional routine method in outpatient PR programs.
2. Determine whether patients who are unable to improve exercise tolerance during conventional exercise training in PR can achieve gains in muscle strength, exercise tolerance, dyspnea, and health status following TCEMS used as an alternate rehabilitative strategy.

ELIGIBILITY:
Inclusion Criteria:

Pulmonary function test criteria consistent with a diagnosis of COPD including forced expiratory volume in one second (FEV1) < 65% of predicted, with FEV1/FVC (forced vital capacity) ratio < 70%, lung hyperinflation based on a residual volume to total lung capacity (RV/TLC) ratio > 120% predicted and reduced diffusing capacity for carbon monoxide (DLCO <70% predicted).

Self-reported exercise limitation despite pharmacologic treatment.

Otherwise medically stable.

Women and minorities will also be recruited. Only persons able to give fully informed consent will be enrolled in the study.

Exclusion Criteria:

Patients will be excluded from study participation if they have a history of uncontrolled cardiovascular disease (including ventricular arrhythmia, myocardial infarction within 1 year, unstable angina, cardiac pacemaker or other implanted electrical device, other uncontrolled arrhythmias, or unstable blood pressure), neuromuscular disease (including stroke), debilitating joint disease or amputations that precludes exercise or have other contraindications to participating in outpatient PR (including unstable bone fracture, syncope of unclear etiology or cancer undergoing active chemotherapy), or are pregnant. Persons with a history of seizure disorder, intracranial clips or skin problems that would prevent safe or proper placement of the electrodes needed for electrical stimulation of the leg muscles will be excluded, based on prior clinical studies of TCEMS in non-COPD populations. Patients will also be excluded from study participation if they have undergone formal PR within 1 year of the date of study inclusion. No patients will be recruited from a "vulnerable patient population", including economically or educationally disadvantaged or mentally disabled persons, children, or prisoners.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2014-05-08 (Actual); Study Completion 2014-05-08 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test (SWT) | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  The incremental Shuttle Walk Test will be used as a measure of exercise capacity. This test measures the maximal distance walked by the patient around two position markers set 10 meters apart, at a pace set by audio signals from a cassette tape. Minute-by-minute walking speed is increased until the patient feels too tired or short of breath to continue, or is unable to walk at least half of the 10 meter distance by the time the next audio signal is heard. Patients who routinely use supplemental oxygen will perform the test while carrying their portable oxygen delivery system during testing. As noted above, a practice run will be performed on the day the patient comes in for familiarization with the protocol and equipment. The investigator conducting the Shuttle Walk Test will be blinded to the groupings of subjects to avoid potential bias of the results.

SECONDARY OUTCOMES:
Body Composition | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  Body composition will be assessed using bioelectrical impedance analysis (Hydra 4200; Xitron Technologies, San Diego, CA) at a standardized time after breakfast. Bioelectrical impedance analysis (BIA) is a simple, safe, non-invasive method to measure assess lean (e.g., muscle) vs. fat body compartments. Fat-free mass will be calculated by using disease-specific equations as described by Schols. Fat mass will then be calculated as total body weight minus fat-free mass. Such BIA measurements are accurate, comparable to other techniques used to assess body composition, and have been validated in patients with COPD.
Body Mass Index (BMI) | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  BMI is calculated as weight in kg/height in m2.
Pulmonary Function | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  Spirometry, lung volume and diffusing capacity measurements will be performed according to standard procedure in the pulmonary function laboratory by a trained pulmonary function technician at either the Newington or West Haven Campus of VACHS according to American Thoracic Society Guidelines.
Muscle Strength | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  Quadriceps and hamstring muscle maximal isokinetic strengths will be measured with the patient in an upright seated position, at an angular velocity of 60 degree/sec using a Biodex Multijoint System 2 dynamometer. Five duplicate leg extension and flexion measurements from a resting knee joint angle of 90 degrees will be made with adequate rest periods (2 min) in between efforts. The best peak torque value in Newton-meter (Nm) unit will be recorded.
Six Minute Walk Test (6MWT) and Borg Dyspnea Rating | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  The total distance walked in 6 minutes is recorded. The 6 minute walk test is well validated for use and is used widely in pulmonary rehabilitation programs, as it is sensitive to changes in exercise endurance that occur following exercise training. The degree of perceived exertion will be assessed at the end of the 6MWT using a Borg Dyspnea scale (a patient-reported numerical rating of the degree of dyspnea associated with any given degree of exertion).
Cardiopulmonary Exercise Test | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  Maximal symptom-limited incremental cardiopulmonary exercise testing (CPET) will be performed by a pulmonary function/exercise technologist according to standard methods used in the West Haven VA Pulmonary Function Laboratory, using a calibrated cycle ergometer (Collins Gold Standard Plus Cardiopulmonary Exercise System, Pulmonary Data Services, Louisville, CO) with a pedaling frequency of 40 revolutions per minute, during which the workload will increase by 5-20 Watt increments every minute depending on the subjects' exercise capacity. Breathing rate, tidal volume, minute ventilation, and electrocardiography will be measured continuously according to standard procedure. Oxygen consumption and carbon dioxide production will be calculated from the fractional concentrations of oxygen and carbon dioxide in the mixed expired gas using a Collins CPX Unit metabolic system (Pulmonary Data Services, Louisville, CO).
Dyspnea Scale | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  The Medical Research Council Dyspnea Scale is a simple questionnaire in which the patient rates the level of exertion/activity at which he/she experiences dyspnea, by checking one of five boxes on a five point scale. This questionnaire takes approximately 5 minutes to complete.
Chronic Respiratory Disease Questionnaire | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  The Chronic Respiratory Disease Questionnaire is a respiratory-specific health status instrument in which patients give responses to simple questions encompassing four principal domains: dyspnea, fatigue, emotion and mastery. This questionnaire is used routinely worldwide as a health status outcomes measure in pulmonary rehabilitation programs, including the outpatient PR program at the West Haven VA, as it is highly responsive to the PR intervention. Total and the four sub-scores for each of the domains tested will be analyzed.
Medical Outcome Survey Short-Form-36 (SF-36) Questionnaire | Baseline, Post 8 Weeks PR, Post 8 Weeks Active/Sham TCEMS
  The SF-36 is a general health status questionnaire in which patients give responses to questions encompassing domains of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Physical and mental summary scores can be calculated from these subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Rochester, MD, Principal Investigator — VA Connecticut Healthcare System/ Yale University School of Medicine
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States